CLINICAL TRIAL: NCT07128771
Title: Cardiomodulatory Effects of Gender-Affirming Hormone Therapy
Acronym: CARMEN
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Collaborators: Oslo University Hospital (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Torbjorn Omland, Professor, University Hospital, Akershus
Other Study IDs: 522599
Record Dates: First submitted 2025-05-30; First posted 2025-08-19 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Gender Incongruence; Cardiovascular Disease (CVD) Risk Factors
Keywords: gender incongruence; gender dysphoria; cardiovascular disease; troponin; NT-proBNP; proteomics; CMR; heart disease; blood pressure; echocardiography; sex hormones; cardiometabolic
MeSH Terms: conditions — Gender Dysphoria; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected at each visit (EDTA-plasma, heparin-plasma and serum).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients receiving gender-affirming hormone therapy: Patients receiving gender-affirming hormone therapy at Oslo University Hospital with a diagnosis of gender-incongruence
- Control group: Age-matched participants not receiving gender-affirming hormone therapy without the diagnosis of gender-incongruence

SUMMARY:
Gender-affirming hormone therapy is today a well-established treatment for individuals experiencing gender-incongruence. However, little is known about the long-term effects of gender-affirming hormone therapy on the cardiovascular system and it is unknown whether gender-affirming hormone therapy is associated with negative, neutral or perhaps positive effects on cardiovascular risk factors. The aim of the study The Cardiomodulatory Effects of Gender-Affirming Hormone Therapy (CARMEN) is therefore to contribute to fill this important knowledge gap by a longitudinal assessment of the affect of gender-affirming hormone therapy with a detailed characterization using state of the art methods for cardiovascular imaging, circulating biomarker assessment, body composition, and self-reported health-related quality of life. The information obtained will inform both candidates for gender-affirming hormone therapy, their families, health personnel and health policy decision makers about the cardiometabolic effects and cardiovascular risks of such therapy and will be relevant information in shared decision-making processes.

DETAILED DESCRIPTION:
The aim of this study is using a prospective and cross-sectional observational design, to assess the effect of initiation and effect of gender-affirming hormone therapy in trans men (female to male) and in trans women (male to female) on:

* Cardiovascular risk factors, including blood pressure, body mass index, body composition, and blood lipids
* Cardiovascular function, structure and anatomy as assessed by cardiovascular magnetic resonance (CMR) imaging and transthoracic echocardiography
* Circulating cardiovascular and inflammatory biomarkers assessed by immunoassays and proteomic profiling
* Self-reported health-related quality of life.

The study will have one longitudinal group where 60 trans women and 60 trans men are followed from the start of treatment till 6-12 months after. An age-matched control group will go through the same assessments.

The second part of the study will be cross-sectional, where the investigators aim to include 100 trans women and 100 trans men already on gender-affirming hormone therapy and being followed at Oslo University Hospital by an endocrinologist.

In both these group, patients who both previously or currently are using Gonadotropin-releasing hormone agonists (GnRH-agonists), so called puberty blockers, will also be eligible for inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gender-incongruence
* Scheduled to initiate gender-affirming hormone therapy at Oslo University Hospital or currently being followed by an endocrinologist for gender-affirming hormone therapy at Oslo University Hospital
* Being 16 years or older

Exclusion Criteria:

- History of clinically significant cardiovascular disease

For the healthy controls, these exclusion criteria also apply:

* No daily smokers
* No endocrine disorders
* No daily medications (except contraception and seasonal medication such as antihistamines)

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients approved for gender-affirming hormone therapy by an endocrinologist at Oslo University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular mass (g) | 6-12 months
  Assessed by cardiac magnetic resonance (CMR) from baseline to end of study.

SECONDARY OUTCOMES:
Change in left ventricular end-systolic volume (LVES) and end-diastolic volume (EDV) (mL) | 6-12 months
  Assessed by cardiac magnetic resonance (CMR) and echocardiography from baseline to end of study.
Change in left ventricle ejection fraction (LVEF) (%) | 6-12 months
  Assessed by cardiac magnetic resonance (CMR) and echocardiography from baseline to end of study.
Change in concentration of circulating cardiac biomarkers | 6-12 months
  Cardiac biomarkers defined as cardiac troponins I and T measured by high sensitivity assays (hs-TnI and hs-TnT) (ng/L) and N-terminal proB-type natriuretic peptide (NT-proBNP) (ng/L), compared from baseline to end of study.
Change in concentration in markers of blood lipids | 6-12 months
  Blood samples will be collected and assessed from baseline to end of study. Blood samples will include markers such as cholesterol, LDL, and HDL (mmol/L).
Change in concentration in markers of cardiometabolic risk factors such as insulin resistance | 6-12 months
  Blood samples will be collected and assessed from baseline to end of study. Blood samples will include the marker HbA1c (mmol/mol).
Changes in global longitudinal strain (GLS) (%) and global circumferential strain (GCS) (%) | 6-12 months
  Assessed by cardiac magnetic resonance (CMR) and echocardiography from baseline to end of study.
Change in arterial stiffness assessed as the pulse wave velocity (m/s) | 6-12 months
  Assessed by cardiac magnetic resonance (CMR) and echocardiography from baseline to end of study.
Change in arterial stiffness assessed as the aortic distensibility (mmHg-1) | 6-12 months
  Assessed by cardiac magnetic resonance (CMR) and echocardiography from baseline to end of study.
Change in blood pressure (mmHg) | 6-12 months
  Blood pressure, both systolic and diastolic blood pressure, will be measured in a standardized manner.
Change in body mass index (BMI) | 6-12 months.
  Weight and height will be measured in a standarized manner and calculated into BMI (kg/m2).
Change in body composition | 6-12 months.
  Body composition will be evaluated using dual-energy x-ray absorptiometry (DXA).
Change in self-reported health-related quality of life (SF-36) | 6-12 months
  For participants aged 18 years or older, the questionnaires SF-36 will be used. SF-36 gives eight scaled scores, each ranging from 0 to 100. Higher scores indicates better health-related quality of life.
Change in self-reported health-related quality of life (PedsQL) | 6-12 months
  For patients aged 16-18, the questionnaire PedsQL will be used. Each question is scored 0-4 and each item response is linearly transformed to a 0-100 scale where higher scores indicate better health-related quality of life.
Change in self-reported health-related quality of life (GHQ-12) | 6-12 months
  For participants aged 18 years or older, the questionnaires GHQ-12 will be used. The scale goes from 0 to 36 (Likert Method) with higher values indicating greater psychological stress.
Change in self-reported health-related quality of life (SDQ) | 6-12 months
  For participants aged 16-18 years of age, the questionnaire SDQ will be used. The scale goes from 0 to 50 with higher values indicating increasing symptoms of difficulties.
Change in self-reported health-related quality of life (Chalders Fatigue Questionnaire) | 6-12 months
  For all participants, the questionnaire Chalders Fatigue Questionnaire will be used. The scale goes from 0 to 33 with higher values indicating increasing symptoms of fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Torbjørn Omland, MD, PhD, MPH, Principal Investigator — University of Oslo
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: No
This is due to data protection considerations.